CLINICAL TRIAL: NCT07176286
Title: An Open-Label, Exploratory, Phase 2 Scintigraphy Study Evaluating 18F-mFBG for Imaging Myocardial Sympathetic Innervation in Subjects With and Without Lewy Body Diseases
Brief Title: 18F-mFBG Cardiac Uptake With Lewy Body Dementia
Acronym: IRP101-231
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Innervate Radiopharmaceuticals LLC (Formerly: Illumina Radiopharmaceuticals LLC) (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: IRP101-231
Record Dates: First submitted 2025-09-10; First posted 2025-09-16 (Actual); Last update posted 2025-10-30 (Actual); Status verified 2025-10

CONDITIONS: Parkinson Disease (PD); Lewy Body Dementia (LBD)
Keywords: IRP101-231; 18F-mFBG
MeSH Terms: conditions — Parkinson Disease; Lewy Body Disease | interventions — 3-fluorobenzylguanidine

STUDY DESIGN:
Intervention Model Description: This is an exploratory study of two study cohorts. Cohort 1 will consist of a minimum of five and maximum of ten participants with known or presumed Lewy body disease (Parkinson's disease (PD) and Lewy body dementia (LBD)). Cohort 2 will consist of participants with neurologic disease due to non-Lewy body pathology.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort 1: Known or presumed Lewy body disease (Parkinson's disease (PD) and Lewy body dementia (LBD) (Active Comparator): All subjects will receive an intravenous injection of 222-370 MBq (6-10 mCi) 18F-mFBG. At 30 minutes post-administration, whole-body imaging will be performed from the head to the pelvis. A static image of the thorax will be acquired at 60 minutes.
  Interventions: Drug: 18F-MFBG
- Cohort 2: neurologic disease due to non-Lewy body pathology. (Active Comparator): All subjects will receive an intravenous injection of 222-370 MBq (6-10 mCi) 18F-mFBG. At 30 minutes post-administration, whole-body imaging will be performed from the head to the pelvis. A static image of the thorax will be acquired at 60 minutes.
  Interventions: Drug: 18F-MFBG

INTERVENTIONS:
Drug: 18F-MFBG — Intravenous injection of 222-370 MBq (6-10 mCi) 18F-mFBG followed by whole body PET imaging.

SUMMARY:
This is a Phase 2 study evaluating the positron-emitting radiopharmaceutical 18F-mFBG as an imaging agent for quantification of the effect of neurodegenerative diseases on myocardial sympathetic innervation. Effectiveness of 18F-mFBG imaging of the heart will be judged in terms of the quantitative difference between results for subjects with Lewy body and non-Lewy body neurologic disease as compared to historical data for healthy control subjects.

DETAILED DESCRIPTION:
Over the past 40 years, significant efforts have been made to develop imaging techniques to monitor the heart's autonomic nervous system, particularly the sympathetic system and its key neurohormone, norepinephrine (NE). In heart disease, NE function is often disrupted, leading to reduced NE uptake and transporter expression, which can contribute to heart failure, arrhythmias, and sudden cardiac death. Similar NE system dysfunction is also seen in neurological conditions like pure autonomic failure (PAF), Parkinson's disease (PD), and Dementia with Lewy Bodies (DLB), which are associated with Lewy body deposits in the nervous system. Most research on myocardial sympathetic neuronal imaging has focused on NE-analogues labeled with gamma- or positron-emitting radioisotopes. The most commonly studied agent is 123I-mIBG, which provides semi-quantitative data. However, its results depend heavily on imaging equipment and techniques, making global standardization difficult. Additionally, accurately measuring myocardial uptake and clearance is challenging with SPECT, even when using correction methods. While most cardiac mIBG research has focused on patients with heart disease, a significant number of studies have examined the effect of Lewy body disease on myocardial sympathetic innervation. These studies have consistently demonstrated a significant reduction in myocardial mIBG uptake. mIBG scintigraphy has high sensitivity (88%) and specificity (85%) for distinguishing Parkinson's disease (PD) from other Parkinsonism disorders. In a study of 123I-mIBG scans, the heart/mediastinum ratio (HMR) showed 68.9% sensitivity and 89.1% specificity for differentiating dementia with Lewy bodies (DLB) from Alzheimer's disease (AD). Neurologists and movement disorder specialists find mIBG imaging helpful for assessing suspected Lewy body disease. Positron-emission tomography (PET) is the preferred method for high-resolution imaging of cellular functions. This study uses 18F-meta-fluorobenzylguanidine (18F-mFBG), a new radiopharmaceutical similar in structure to 123I-mIBG but with faster pharmacokinetics and elimination. Compared to 123I-mIBG, 18F-mFBG clears more quickly from the blood and target organs, resulting in better heart imaging quality and reliability. While most research on 18F-mFBG has focused on imaging neural crest tumors like neuroblastoma and pheochromocytoma, its performance is expected to be strong based on prior experience with 123I-mIBG. With the greater sensitivity and resolution of PET imaging compared to planar and SPECT techniques, it is expected that 18F-mFBG imaging will be less procedure-dependent than 123I-mIBG and provide the reliable and reproducible quantitative accuracy necessary to support use of this agent for clinical patient studies.

ELIGIBILITY:
Inclusion Criteria:

* 1. ≥18 years of age at study entry. 2. Able and willing to comply with study procedures and signed and dated informed consent is obtained.

  3. A male or a female who is either surgically sterile (has had a documented bilateral oophorectomy and/or hysterectomy), postmenopausal (cessation of menses for more than 1 year), non-lactating, or of childbearing potential for whom the result of a serum pregnancy test performed at screening is negative.

  4. All subjects: Judged clinically stable for at least 30 days before enrolment into the study and remains stable to the time of the study imaging procedure.

For Lewy body disease subjects (Study Cohort I):

5. The subject has a diagnosis of either PD or DLB based on accepted clinical criteria at least 6 months before enrollment into the study.

For non-Lewy body disease subjects (Study Cohort II):

6. The subject has a diagnosis of neurological or neurodegenerative disease for which neither PD nor DLB is judged likely by a neurologist based on accepted clinical and imaging criteria.

Exclusion Criteria:

* 1. Previously entered into this study or has participated in any other investigational product or medical device study within 30 days of enrollment.

  2. History or suspicion of significant allergic reaction or anaphylaxis to any components of the 18F-mFBG imaging agent.

  3. Presents with any other clinically active, serious, life-threatening disease with a life expectancy of less than 1 year or where participation in the study might compromise the management of the subject or other reason that in the judgment of the investigator(s) makes the subject unsuitable for participation in the study.

  4. Documented ischemic heart disease (prior myocardial infarction, unstable angina, etc) or a diagnosis of heart failure of ischemic or non-ischemic etiology.

  5. Serious non-cardiac medical condition associated with significant elevation of plasma catecholamines including pheochromocytoma.

  6. The subject is claustrophobic or has a movement disorder that prevents him/her from lying still in a supine position for up to 20 minutes.

  7. Renal insufficiency (serum creatinine >3.0 mg/dL). 8. Uses medications that are known to interfere with uptake of NET-dependent agents and these medications cannot be safely withheld 24 hours before study procedures.

  9. Participated in a research study using ionizing radiation in the previous 12 months such that participation in the study might result in a total effective dose from research procedures exceeding 50 milliSieverts during that time interval.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-11-30 (Estimated); Primary Completion 2026-05-30 (Estimated); Study Completion 2026-07-30 (Estimated)

PRIMARY OUTCOMES:
Cohort 1: Quantify the extent and degree of global and regional reduced 18F-mFBG myocardial uptake on PET/CT (or PET/MR) of subjects with known or presumed Lewy body disease (Parkinson's disease (PD) and Lewy body dementia (LBD)). | 6 months
  All image data will be analyzed to develop and validate quantitative measures of global and regional myocardial uptake of 18F-mFBG at two times between injection and 60 minutes post-administration. The data from subjects without Lewy body disease will be used in comparisons with equivalent results for Lewy body disease subjects. Results for subjects imaged in this study will also be compared with historical data from imaging of healthy control subjects without heart disease.

SECONDARY OUTCOMES:
Cohorts 1 and 2: Quantify 18F-mFBG whole-body activity distribution in Lewy body disease subjects (voxel, regional, and global basis) at 30-minutes post-administration | 6 months
  Normalized uptake measurements (counts/voxel/MBq administered) determined from Lewy body disease subjects will be used for quantitative comparisons to non-Lewy body disease and historical healthy control subject scans.
Cohort 1 and 2: 18F-mFBG PET quantitative assessment at 60 minutes | 6 months
  18F-mFBG myocardial activity in Lewy body disease subjects (voxel, regional, and global basis) at 60-minutes post-administration compared to non-Lewy body disease subjects.
Cohorts 1 and 2: Global myocardial 18F-mFBG activity in Lewy body disease subjects compared to non-Lewy body disease subjects. | 6 months
  Global myocardial 18F-mFBG activity in Lewy body disease subjects at 30-minutes post-administration, as a proportion of total-body activity, compared to non-Lewy body disease subjects.

CONTACTS AND LOCATIONS:
Overall Officials: Juan B Toledo, MD, Principal Investigator — The Methodist Hospital Research Institute

IPD SHARING:
Plan to Share IPD: No